CLINICAL TRIAL: NCT06089226
Title: The Relationship Between Physical Activity Level and Cardiovascular Fitness and Respiratory Parameters in Individuals With Spinal Cord Injury
Brief Title: Parameters Related to Physical Activity Level in SCI
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Kubra Koce, Lecturer, Istinye University
Other Study IDs: 23/198
Record Dates: First submitted 2023-09-20; First posted 2023-10-18 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injuries; Respiratory Complication; Cardiovascular Complication
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assessment Group
  Interventions: Other: Assessment Group

INTERVENTIONS:
Other: Assessment Group — In our prospectively planned study, patients who meet the inclusion criteria will be evaluated by the researcher via face-to-face interview method and the evaluations specified in the outcome measurements. Patients participating in the study will first be given a general explanation about the purpose of the study and evaluation methods, and their written consent will be obtained.

SUMMARY:
Spinal cord injury (SCI) is a devastating health condition associated with permanent disability and reduced life expectancy. It is stated that its annual incidence worldwide varies between 12.1 and 57.8 per million, and its prevalence varies between 236 and 1009 per million.

SCI negatively affects the physical, psychological, and social well-being of individuals by causing sensory, motor, and autonomic dysfunction. The level of disability associated with SCI is different for each injury and varies depending on the level and type of injury. However, physical activity (PA), cardiovascular fitness, and respiratory system are commonly observed to be affected in most individuals with SCI.

Due to inadequate control of somatic and autonomic systems, a decrease in the cardiovascular response to PA and exercise occurs. A decrease in PA level and systemic disorders after injury promote sedentary behavior and negatively affect cardiovascular fitness in individuals with SCI. Cervical and thoracic spinal cord injuries compromise the function of the respiratory muscles and significantly impair both inspiratory and expiratory function. It also interrupts the sympathetic innervation of the lungs and creates restrictive changes in the physiological and mechanical properties of the lungs. The broad effects of SCI on lung capacity may have implications for cardiovascular fitness. Adequate ventilation is critical to provide adequate oxygen to working muscles during prolonged physical activities. During moderate and high-intensity physical activities, ventilation increases in proportion to oxygen consumption to maintain arterial oxygen concentration and allow continuous PA.

Knowing the relationship between PA, cardiovascular fitness, and respiratory parameters after SCI is essential in guiding the course of rehabilitation after SCI. Battikha et al. They reported that respiratory capacity plays an important role in limiting exercise capacity in individuals with SCI. However, the relationship between PA and cardiovascular fitness and respiratory parameters has not been fully examined in individuals with SCI.

In this study, the investigators hypothesize the relationship between PA, cardiovascular fitness and respiratory parameters. Accordingly, this study aims to determine the relationship between PA, cardiovascular fitness and respiratory parameters in individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Classified as group A, B, C or D (diagnosed with spinal cord injury) according to the American Spinal Injury Association (ASIA),
* Fully or partially wheelchair dependent
* Having the upper extremity muscle strength required to use a wheelchair
* Those who are over 18 years old
* Patients without cognitive impairment

Exclusion Criteria:

* Those with any progressive disease
* Bedridden,
* Patients with severe cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with spinal cord injury classified as group A, B, C or D according to the American Spinal Injury Association (ASIA)
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity Scale for Individuals with Physical Disabilities | 1 week
  Physical Activity Scale for Individuals with Physical Disabilities will be used to evaluate the physical activity level of individuals with SCI. The scale is a 13-item self-report form for classification purposes covering daily living activities (items 1-6), domestic activities (items 7-12) and professional duties (item 13) in the last seven days.A high score indicates a high level of physical activity.
The Wheelchair Propulsion Test | 1 week
  It will be used to evaluate the cardiovascular fitness level of participants. The test includes a total of 3 tests: 20 Meter Propulsion Test, Slalom Test and 6 Minute Push Test. In the 20 Meter Propulsion Test, the number of seconds in which the participant completes 20 meters is measured with a stopwatch. A high value indicates low cardiovascular fitness. In the Slalom Test, the number of seconds in which the participant completes the 8-way track is measured with a stopwatch. A high value indicates low cardiovascular fitness. In the 6-minute push test, the distance traveled by the participant during 6 minutes is measured in meters. A higher value indicates higher cardiovascular fitness.
Forced vital capacity | 1 week
  Forced vital capacity is the volume of gas expelled from the lungs in a fast, forced and deep expiration after a deep, forced inspiration. Forced vital capacity will be performed in a sitting position using a portable spirometer (Spirobank; MIR, Rome, Italy) according to American Thoracic Society guidelines.
Forced expiratory volume in the first second | 1 week
  Forced expiratory volume in the first second is the amount of air expelled from the lungs in the first second with forced expiration. Forced expiratory volume in the first second will be performed in a sitting position using a portable spirometer (Spirobank; MIR, Rome, Italy) according to American Thoracic Society guidelines.
Forced vital capacity/Forced expiratory volume Ratio | 1 week
  The Forced vital capacity/Forced expiratory volume Ratio, also called the modified Tiffeneau-Pinelli index, is a calculated ratio used in the diagnosis of obstructive and restrictive lung disease. The ratio will be performed in a sitting position using a portable spirometer (Spirobank; MIR, Rome, Italy) according to American Thoracic Society guidelines.
Peak expiratory flow rat | 1 week
  Peak expiratory flow rate is the volume of air forcefully expelled from the lungs in one quick exhalation, and is a reliable indicator of ventilation adequacy as well as airflow obstruction. The ratio will be performed in a sitting position using a portable spirometer (Spirobank; MIR, Rome, Italy) according to American Thoracic Society guidelines.
Respiratory muscle strength | 1 week
  Respiratory muscle strength, maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be assessed using an electronic pressure transducer (MicroRPM; Micro Medical Ltd., Kent, United Kingdom).

SECONDARY OUTCOMES:
Sociodemographic Information and Health Status Information | 4 weeks
  Participants' sociodemographic information and health status information will be recorded in the Patient Evaluation Form. The Patient Evaluation Form prepared by the researcher consists of 2 parts. First part; It consists of 15 questions that include information such as the patient's age, gender, height, weight, profession, and educational status. The second part consists of 7 questions containing information such as the cause of injury, ASIA level, neurological injury level, and ambulation level. The answers received from the patients will be recorded in the evaluation form.
Body Weight Measurement | 1 week
  It is a measure that shows the sum of body weight, fat mass and fat-free mass, and is used quite often because it is practical.The body weights of the participants, as described in the literature, will initially be weighed with an electronic scale while they are dressed and sitting in a wheelchair, and then the wheelchair and their clothes will be weighed and subtracted from the total weight. The result will be recorded on the evaluation form in kilograms.
Height Measurement | 1 week
  The height of the participants will be measured with a non-stretchable tape measure as described in the literature, in the supine position, the head in the Frankfort position, the legs stretched, and the feet in dorsiflexion, and the result will be recorded in the evaluation form in centimeters.
Body mass index | 1 week
  Body mass index will be calculated as weight (kg) / height² (cm²) and recorded in the evaluation form.
Waist Circumference Measurement | 1 week
  An easier way to evaluate obesity in individuals with spinal cord injury is waist circumference measurement, which gives an idea about body fat distribution rather than total fat amount. Participants' waist circumferences will be measured with a non-flexible tape measure at the end of normal expiration, with their clothes removed and their arms at their sides, and recorded in centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided